CLINICAL TRIAL: NCT04514068
Title: Effect of Electroacupuncture on P6 Acupoint on Hypertensive Patients.
Acronym: EEP6
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ong Fujian Chinese Physician Hall (Other)
Responsible Party: Principal Investigator, Lin Ho Wong, Director, Ong Fujian Chinese Physician Hall
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OngFujianCPH
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
Keywords: acupuncture
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unilateral electroacupuncture of p6 acupoint (Experimental)
  Interventions: Procedure: Acupuncture
- Bilateral electroacupuncture of p6 acupoint (Experimental)
  Interventions: Procedure: Acupuncture
- Sham acupuncture of p6 acupoint (Sham Comparator)
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — In each session, acupuncture are applied unilaterally or bilaterally on P6 acupoint. Each acupuncture needle will be stimulated by transcutaneous electric device.
  Arms: Bilateral electroacupuncture of p6 acupoint; Unilateral electroacupuncture of p6 acupoint
Procedure: Sham acupuncture — Sham acupuncture
  Arms: Sham acupuncture of p6 acupoint

SUMMARY:
This is a randomized controlled clinical trial with three parallel arms. This trial aims to evaluate the effectiveness of electroacupuncture on P6 acupoint for patients with hypertension,with respect to decreasing their blood pressure, safety of acupuncture ,and improving their quality of life as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old
* Have not recently had any changes in anti-hypertensive medications
* Have not recently been discharged from hospital/are stable
* Is not having any acute infection.

Exclusion Criteria:

* Trypanophobia
* Below 18 years of age
* Is currently having an acute infection
* Is unstable or have been discharged recently from hospital
* Changes made to anti-hypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of blood pressure. | up to 6 months
  It is expected that both blood pressure and heart rate will be reduced during the electroacupuncture of P6 acupoint.
Reduction of Heart Rate | up to 6 months
  Heart Rate is also expected to be reduced with the stimulation of p6 acupoint.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ho Wong, MB BCH BAO, Study Director — Ong Fujian Chinese Physician Hall; Pang Ong Wong, PhD, Principal Investigator — Ong Fujian Chinese Physician Hall; Eng Soon Ong, Bachelor of TCM, Study Chair — Ong Fujian Chinese Physician Hall; Choo Keok Lim, PhD, Study Chair — Ong Fujian Chinese Physician Hall
Locations (1):
- Ong Fujian Chinese Physician Hall, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No